CLINICAL TRIAL: NCT02193139
Title: A Randomized, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of An Anticholinergic Agent for the Treatment of Primary Axillary Hyperhidrosis
Brief Title: Safety and Efficacy of an Anticholinergic Agent for Treatment of Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OH1304
Record Dates: First submitted 2014-06-29; First posted 2014-07-17 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2014-11

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- WL8713, 6 mg (Experimental): 6 mg WL8713 administered daily
  Interventions: Drug: WL8713, 6 mg
- WL8713, 12 mg (Experimental): 12 mg WL8713 administered daily
  Interventions: Drug: WL8713, 12 mg
- WL8713, 18 mg (Experimental): 18 mg WL8713 administered daily
  Interventions: Drug: WL8713, 18 mg
- WL8713, 24 mg (Experimental): 24 mg WL8713 administered daily
  Interventions: Drug: WL8713, 24 mg
- Placebo (Placebo Comparator): placebo administered daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WL8713, 6 mg
  Arms: WL8713, 6 mg
Drug: WL8713, 12 mg
  Arms: WL8713, 12 mg
Drug: WL8713, 18 mg
  Arms: WL8713, 18 mg
Drug: WL8713, 24 mg
  Arms: WL8713, 24 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Phase 2 study is designed to evaluate multiple doses of an anticholinergic-containing medication and identify the dose or doses that may effectively reduce axillary sweating in hyperhidrotic subjects. The anticholinergic agent being studied is designated WL8713.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with primary axillary hyperhidrosis
* Poor quality of life rating on the Hyperhidrosis Disease Severity Scale (score of 3 or 4)
* Has a baseline gravimetric measurement of spontaneous resting sweat production of ≥100 mg/10 min at room at room temperature in at least one axilla
* Meets at least two of the following criteria (self-reported):

  * sweating is bilateral and symmetrical
  * excessive sweating impairs daily activities
  * subject experiences at least one sweating episode per week
  * excessive sweating onset was earlier than age 25 years
  * has a positive family history for excessive sweating
  * cessation of sweating during sleep

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Gravimetric measurement of sweat production | 6 weeks
  Change from baseline in mean (bilateral average) sweat weight at Week 6 (LOCF)

SECONDARY OUTCOMES:
Hyperhidrosis Disease Severity Scale (HDSS) scores | 6 weeks
  Percentage of subjects with a change from baseline in HDSS scores of at least -2 points at Week 6 (LOCF)
Dermatology Life Quality Index (DLQI) scores | 6 weeks
  Change from baseline in DLQI total score at Week 6 (LOCF)
Global Assessment of Disease State responses | 6 weeks
  Global Assessment of Disease State score at Week 6 (LOCF)

CONTACTS AND LOCATIONS:
Locations (1):
- Watson Clinical Site, San Diego, California, United States